CLINICAL TRIAL: NCT02246413
Title: RCT on Co-management of Obesity, Depression, and Elevated CVD Risk in Primary Care-- Engaging Self-regulation Targets to Understand the Mechanisms of Behavior Change and Improve Mood and Weight Outcomes
Brief Title: Research Aimed at Improving Both Mood and Weight
Acronym: RAINBOW-ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Washington (Other); University of Pittsburgh (Other); Stanford University (Other); University of Illinois at Chicago (Other); Sutter Health (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, PhD, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 14-05-323; R01HL119453 (NIH); UH2HL132368 (NIH)
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Depression; Obesity
Keywords: BMI; Depressive symptoms; Integrated therapy; Cardiometabolic risk; Self-regulation; Behavior change; Precision medicine; Lifestyle
MeSH Terms: conditions — Depression; Obesity; Self-Control

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAINBOW Intervention Program (Experimental): An integrated intervention program for helping to improve mood and weight in adults who may be at risk for diabetes and heart disease.
  Interventions: Behavioral: RAINBOW Intervention Program
- Usual Care (No Intervention): Usual Care.

INTERVENTIONS:
Behavioral: RAINBOW Intervention Program — Integrated lifestyle intervention with as-needed antidepressant pharmacotherapy to treat coexisting obesity and depression in adults in primary care
  Arms: RAINBOW Intervention Program

SUMMARY:
The RAINBOW study is an NIH R01-funded randomized controlled trial to evaluate the clinical and cost effectiveness and implementation potential of a primary care integrated multicondition intervention program to help improve mood and weight for obese adults with clinically significant depressive symptoms. The ENGAGE study is a mechanistic investigation added to the main trial with funding through the NIH common fund for the Science of Behavior Change roadmap initiative. Beginning Jan 11, 2016, at least 100 of newly enrolled trial participants will be consented to undergo additional assays evaluating neurobiological mechanisms of self-regulation.

DETAILED DESCRIPTION:
The large numbers of primary care patients affected by coexisting obesity and depression and common risk factors for diabetes and heart disease underscore the urgency of developing effective, accessible, and sustainable interventions that use an integrated, multicondition care management approach. The RAINBOW trial will rigorously evaluate the clinical and cost effectiveness and potential for "real-world" implementation of an innovative intervention that integrates a behavioral weight loss program and a collaborative stepped care program for depression, incorporates conventional clinic- and home-based modes of care delivery (e.g., office visits plus phone consults and take-home DVD), and leverages low-cost, wide-reach health information technologies (e.g., Web, secure email, and mobile texting). Beginning Jan 11, 2016, at least 100 of newly enrolled trial participants will also be consented to undergo additional assays evaluating neurobiological mechanisms of self-regulation, including emotional regulation, cognitive control and self-reflection. Given its focus on transforming primary care management of obesity and depression and common cardiometabolic risk factors to evidence-based, patient-centered care, as well as the likely scalability of the proposed intervention, the study has high potential for significant clinical and public health impact. Furthermore, elucidating the neurobiological mechanisms of self-regulation will significantly advance precision lifestyle medicine by enabling mechanism-targeted individualization of treatment.

ELIGIBILITY:
RAINBOW

Inclusion criteria:

* Ethnicity and race: Any;
* Obesity: BMI≥30 kg/m2 for non-Asians; BMI≥27 kg/m2 for Asians;
* Clinically significant depressive symptoms: PHQ-9≥10;
* A PAMF patient for ≥1 year
* Seen in primary care at least once in the preceding 24 months;
* Able and willing to enroll and meet the requirements of the study

Exclusion criteria:

* Inability to speak, read or understand English;
* Having no reliable telephone service, no device to use to watch a DVD, or no regular Internet access via a computer and/or mobile device;
* Had bariatric surgery within the past 12 months or plans to undergo bariatric surgery during the 24-month study period;
* Ongoing psychiatric care outside of the PAMF network.
* Active suicidal ideation that includes active plan and/or intent;
* Any Axis I disorder other than Minor or Major Depressive Disorder and/or Dysthymia, with the exception of any comorbid Anxiety Disorder;
* Active Bulimia Nervosa within the past 12 months (however Binge Eating Disorder without purging is not an exclusionary condition);
* Active alcohol or substance use disorder (including prescription drugs).
* Pre-existing diabetes (other than during pregnancy) or diabetes diagnosed as a result of fasting blood glucose or hemoglobin A1c levels obtained through study screening;
* Pre-existing cardiovascular disease.
* Diagnosis of cancer (other than non-melanoma skin cancer) that is/was active or treated with radiation or chemotherapy within the past 12 months;
* Severe medical comorbidities that require aggressive treatment, e.g., stage 4 or greater renal disease, liver failure;
* Diagnosis of a terminal illness and/or in hospice care;
* Residence in long-term care facility;
* Cognitive impairment based on the Callahan 6-item scale
* Plan to move out of the area or transfer care outside PAMF during the study period;
* Investigator discretion for reasons of clinical safety or protocol adherence.

ENGAGE

Inclusion criteria:

• RAINBOW participant

Exclusion criteria:

* Weight over 350 pounds
* MRI is contraindicated
* Traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, PhD, Principal Investigator — University of Illinois at Chicago; Leanne Williams, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Palo Alto Medical Foundation, Palo Alto, California
  - Stanford University, Stanford, California

REFERENCES:
- [Derived] Lv N, Chin SW, Xiao L, Tang Z, Parikh A, Ma J. Sex moderates diet quality differences in integrated collaborative care for comorbid obesity and depression: Post-hoc analysis of the RAINBOW RCT. J Nutr Health Aging. 2025 Jan;29(1):100426. doi: 10.1016/j.jnha.2024.100426. Epub 2024 Nov 29. PMID 39615398
- [Derived] Zhang X, Pines A, Stetz P, Goldstein-Piekarski AN, Xiao L, Lv N, Tozzi L, Lavori PW, Snowden MB, Venditti EM, Smyth JM, Suppes T, Ajilore O, Ma J, Williams LM. Adaptive cognitive control circuit changes associated with problem-solving ability and depression symptom outcomes over 24 months. Sci Transl Med. 2024 Sep 4;16(763):eadh3172. doi: 10.1126/scitranslmed.adh3172. Epub 2024 Sep 4. PMID 39231241
- [Derived] Kannampallil T, Dai R, Lv N, Xiao L, Lu C, Ajilore OA, Snowden MB, Venditti EM, Williams LM, Kringle EA, Ma J. Cross-trial prediction of depression remission using problem-solving therapy: A machine learning approach. J Affect Disord. 2022 Jul 1;308:89-97. doi: 10.1016/j.jad.2022.04.015. Epub 2022 Apr 7. PMID 35398399
- [Derived] Lv N, Lefferts WK, Xiao L, Goldstein-Piekarski AN, Wielgosz J, Lavori PW, Simmons JM, Smyth JM, Stetz P, Venditti EM, Lewis MA, Rosas LG, Snowden MB, Ajilore OA, Suppes T, Williams LM, Ma J. Problem-solving therapy-induced amygdala engagement mediates lifestyle behavior change in obesity with comorbid depression: a randomized proof-of-mechanism trial. Am J Clin Nutr. 2021 Dec 1;114(6):2060-2073. doi: 10.1093/ajcn/nqab280. PMID 34476464
- [Derived] Goldstein-Piekarski AN, Wielgosz J, Xiao L, Stetz P, Correa CG, Chang SE, Lv N, Rosas LG, Lavori PW, Snowden MB, Venditti EM, Simmons JM, Smyth JM, Suppes T, Lewis MA, Ajilore O, Ma J, Williams LM. Early changes in neural circuit function engaged by negative emotion and modified by behavioural intervention are associated with depression and problem-solving outcomes: A report from the ENGAGE randomized controlled trial. EBioMedicine. 2021 May;67:103387. doi: 10.1016/j.ebiom.2021.103387. Epub 2021 May 17. PMID 34004422
- [Derived] Lv N, Xiao L, Rosas LG, Venditti EM, Smyth JM, Lewis MA, Snowden MB, Ronneberg CR, Williams LM, Gerber BS, Ajilore OA, Patel AS, Ma J. Sex Moderates Treatment Effects of Integrated Collaborative Care for Comorbid Obesity and Depression: The RAINBOW RCT. Ann Behav Med. 2021 Nov 18;55(12):1157-1167. doi: 10.1093/abm/kaaa125. PMID 33616188
- [Derived] Goldhaber-Fiebert JD, Prince L, Xiao L, Lv N, Rosas LG, Venditti EM, Lewis MA, Snowden MB, Ma J. First-Year Economic and Quality of Life Effects of the RAINBOW Intervention to Treat Comorbid Obesity and Depression. Obesity (Silver Spring). 2020 Jun;28(6):1031-1039. doi: 10.1002/oby.22805. Epub 2020 Apr 22. PMID 32320533
- [Derived] Lv N, Xiao L, Majd M, Lavori PW, Smyth JM, Rosas LG, Venditti EM, Snowden MB, Lewis MA, Ward E, Lesser L, Williams LM, Azar KMJ, Ma J. Variability in engagement and progress in efficacious integrated collaborative care for primary care patients with obesity and depression: Within-treatment analysis in the RAINBOW trial. PLoS One. 2020 Apr 21;15(4):e0231743. doi: 10.1371/journal.pone.0231743. eCollection 2020. PMID 32315362
- [Derived] Rosas LG, Azar KMJ, Lv N, Xiao L, Goldhaber-Fiebert JD, Snowden MB, Venditti EM, Lewis MM, Goldstein-Piekarski AN, Ma J. Effect of an Intervention for Obesity and Depression on Patient-Centered Outcomes: An RCT. Am J Prev Med. 2020 Apr;58(4):496-505. doi: 10.1016/j.amepre.2019.11.005. Epub 2020 Feb 14. PMID 32067873
- [Derived] Ma J, Rosas LG, Lv N, Xiao L, Snowden MB, Venditti EM, Lewis MA, Goldhaber-Fiebert JD, Lavori PW. Effect of Integrated Behavioral Weight Loss Treatment and Problem-Solving Therapy on Body Mass Index and Depressive Symptoms Among Patients With Obesity and Depression: The RAINBOW Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):869-879. doi: 10.1001/jama.2019.0557. PMID 30835308
- [Derived] Ma J, Xiao L, Lv N, Rosas LG, Lewis MA, Goldhaber-Fiebert JD, Venditti EM, Snowden MB, Lesser L, Ward E. Profiles of sociodemographic, behavioral, clinical and psychosocial characteristics among primary care patients with comorbid obesity and depression. Prev Med Rep. 2017 Aug 5;8:42-50. doi: 10.1016/j.pmedr.2017.07.010. eCollection 2017 Dec. PMID 28840096
- [Derived] Ma J, Yank V, Lv N, Goldhaber-Fiebert JD, Lewis MA, Kramer MK, Snowden MB, Rosas LG, Xiao L, Blonstein AC. Research aimed at improving both mood and weight (RAINBOW) in primary care: A type 1 hybrid design randomized controlled trial. Contemp Clin Trials. 2015 Jul;43:260-78. doi: 10.1016/j.cct.2015.06.010. Epub 2015 Jun 19. PMID 26096714

RESULTS

PARTICIPANT FLOW:
Period: 12-months (Primary Outcome)
Arm/Group | RAINBOW Intervention Program | Usual Care
Started | 204 | 205
Completed | 169 | 175
Not Completed | 35 | 30
Period: 24-months (Secondary Outcome)
Arm/Group | RAINBOW Intervention Program | Usual Care
Started | 204 | 205
Completed | 153 | 173
Not Completed | 51 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAINBOW Intervention Program | Usual Care | Total
Number analyzed (Participants) | 204 | 205 | 409
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (12.2) | 51.0 (11.9) | 51.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 143 | 287
  Male | 60 | 62 | 122
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 147 | 142 | 289
  African American | 3 | 3 | 6
  Asian/Pacific Islander | 20 | 20 | 40
  Hispanic | 26 | 30 | 56
  Other | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 204 | 205 | 409
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: 287 women plus 122 men equal to the 409 total sample.
  kg/m^2
    All | 36.7 (6.9) | 36.6 (5.8) | 36.7 (6.4)
    Women: number analyzed (Participants) | 144 | 143 | 287
    Women | 36.8 (6.6) | 37.3 (5.9) | 37.0 (6.2)
    Men: number analyzed (Participants) | 60 | 62 | 122
    Men | 36.4 (7.5) | 35.1 (5.5) | 35.7 (6.6)
Patient Health Questionnaire 9-items (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The 9-item Patient Health Questionnaire (PHQ-9) total score is the sum of the scores of the 9 items, ranging from 0 to 27. Higher scores represent more severe depression symptoms. Scores of 5, 10, 15, and 20 represent cut points for mild, moderate, moderately severe and severe depression, respectively.
  units on a scale | 14.1 (3.2) | 13.5 (3.0) | 13.8 (3.1)
Depression Symptom Checklist 20-items (SCL-20) [Mean (Standard Deviation); unit: units on a scale] — Depression Symptom Checklist 20 (SCL-20), total average scores of the 20 items with a range from 0 (not at all) to 4 (extremely). Higher scores represent more severe depression symptoms. SCL-20 cutoff points of 1.5 and 2.0 correspond to moderate and severe depression, respectively.
  units on a scale | 1.5 (0.5) | 1.5 (0.6) | 1.5 (0.5)
Taking antidepressant medications [Count of Participants; unit: Participants] | 85 | 84 | 169

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Outcome: Body Mass Index (BMI)
Description: Integrated intervention treatment response
Time Frame: 12 months
Population: In the case of missing study-measured weight, the closest EHR weight within 3 months of the due date of a missed study visit or self-reported weight (if no EHR weight) was used. So the number of participants analyzed is not consistent with the number in the Participant Flow module.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 183 | 184
kg/m^2 | 35.9 (7.1) | 36.6 (6.0)

2. Primary Outcome: Co-Primary Outcome: Depression Symptom Checklist 20 (SCL-20) Score
Description: Depression Symptom Checklist 20 (SCL-20) questionnaire score. SCL-20, average scores of the 20 items with a range from 0 (not at all) to 4 (extremely). SCL-20 cutoff points scores of ≤0.75, >0.75-1.5, >1.5- 2.0, and >2.0 represent remission, mild depression, moderate depression, and severe depression, respectively.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 169 | 175
score on a scale | 1.1 (0.7) | 1.4 (0.9)

3. Secondary Outcome: Body Mass Index
Description: Derived from height and weight measurements
Time Frame: 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 178 | 179
kg/m2 | 36.2 (7.3) | 36.2 (6.5)

4. Secondary Outcome: Depression Symptom Checklist 20 (SCL-20) Score
Description: SCL-20 full questionnaire. SCL-20, average scores of the 20 items with a range from 0 (not at all) to 4 (extremely). SCL-20 cutoff points scores of ≤0.75, >0.75-1.5, >1.5- 2.0, and >2.0 represent remission, mild depression, moderate depression, and severe depression, respectively.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 153 | 173
score on a scale | 1.3 (0.8) | 1.4 (0.9)

5. Secondary Outcome: Weight
Description: Weight measurements
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 183 | 184
kg | 100.8 (22.8) | 103.4 (20.9)

6. Secondary Outcome: Weight
Description: Weight measurements
Time Frame: 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 178 | 179
kg | 101.8 (24) | 102.4 (22.4)

7. Secondary Outcome: Depression Remission (Number of Participants With SCL-20 Scores <0.5)
Description: Depression remission defined by Depression Symptom Checklist 20 (SCL-20) scores <0.5
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 169 | 175
Participants | 30 | 23

8. Secondary Outcome: Depression Remission (Number of Participants With SCL-20 Score <0.5)
Description: Depression remission defined by Depression Symptom Checklist 20 (SCL-20) scores <0.5
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 153 | 173
Participants | 31 | 20

9. Secondary Outcome: Depression Treatment Response (Number of Participants With ≥50% Decrease in SCL-20 Scores From Baseline)
Description: Depression treatment response defined by 50% decline in SCL-20 symptom scores
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 169 | 175
Participants | 49 | 38

10. Secondary Outcome: Depression Treatment Response (Number of Participants With ≥50% Decrease in SCL-20 Scores From Baseline)
Description: Depression treatment response defined by 50% decline in SCL-20 symptom scores
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 153 | 173
Participants | 40 | 39

11. Secondary Outcome: Clinically Significant Weight Loss (Number of Participants With ≥5% Weight Loss From Baseline)
Description: 5% or greater weight loss from baseline
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 183 | 184
Participants | 51 | 27

12. Secondary Outcome: Clinically Significant Weight Loss (Number of Participants With ≥5% Weight Loss From Baseline)
Description: 5% or greater weight loss from baseline
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 178 | 179
Participants | 42 | 37

13. Secondary Outcome: Cost-effectiveness
Description: Average annual per person spending on medical care services (2018 real US dollars)
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: US dollars
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 178 | 180
US dollars | 1994 [1473 to 2515] | 1773 [1209 to 2337]

14. Secondary Outcome: Obesity-related Psychosocial Functioning (Obesity-related Problem Scale)
Description: Obesity-related Problem Scale, average scores of 8 questions with a range from 0 (no at all) to 3 (extremely). The average score is then multiplied by 100 and divided by 3 to convert to a scale of 0-100, with a higher score indicating more obesity-related problems.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 137
score on a scale | 54.3 (25.9) | 56.1 (27.2)

15. Secondary Outcome: Anxiety (GAD-7)
Description: Self-administered questionnaire. Total scores of the 7 items with a range from 0 (no symptoms) to 21 (most severe symptoms).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 131 | 137
score on a scale | 4.6 (3.8) | 6.1 (4.6)

16. Secondary Outcome: Generic Health-related Quality of Life (SF-8 - Physical Component (PCS) )
Description: Self-administered questionnaire - Generic Health-related Quality of Life (SF-8 - physical component (PCS) ) Physical and mental composite scores, a population scale ranged from 0 (lowest quality of life) to 100 (highest quality of life) summed by the total converted scores of each value of the 8 questions. These summary scales have been normalized in the U.S. population (value=50). The higher score indicates better self-reported health-related quality of life.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 138
score on a scale | 47.1 (8.7) | 46.3 (8.6)

17. Secondary Outcome: Generic Health-related Quality of Life (SF-8 - Mental Component (MCS) )
Description: Self-administered questionnaire - Generic Health-related Quality of Life (SF-8 - Mental Component (MCS) ). Physical and mental composite scores, a population scale ranged from 0 (lowest quality of life) to 100 (highest quality of life) summed by the total converted scores of each value of the 8 questions. These summary scales have been normalized in the U.S. population (value=50). The higher score indicates better self-reported health-related quality of life.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 138
score on a scale | 45 (9.6) | 43.3 (9.5)

18. Secondary Outcome: Disability (Sheehan Disability Scale)
Description: Self-administered Sheehan Disability Scale questionnaire. Sheehan Disability Scale, total scores of the 3 items with a range from 0 (unimpaired) to 30 (highly impaired). Scores of ≥5 on any of the 3 scales (Work/school [0-10], Social life [0-10], and Family life/home responsibilities [0-10]) are associated with signiﬁcant functional impairment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 129 | 132
score on a scale | 6.8 (6.7) | 8.4 (6.2)

19. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Activity)
Description: Self-administered questionnaire: Utility-based Health-related Quality of Life - USUAL ACTIVITIES (e.g. work, study, housework, family or leisure activities). A 5-point scale (1) No problems, (2) Slight problems, (3) Moderate problems, (4) Severe problems, and (5) Extreme problems.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 138
score on a scale | 1.4 (0.7) | 1.6 (0.8)

20. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Pain)
Description: Self-administered questionnaire: Utility-based Health-related Quality of Life - PAIN/DISCOMFORT. A 5-point scale (1) No problems, (2) Slight problems, (3) Moderate problems, (4) Severe problems, and (5) Extreme problems.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 138
score on a scale | 2.0 (0.8) | 2.1 (0.8)

21. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Anxiety/Depression)
Description: Self-administered questionnaire: Utility-based Health-related Quality of Life - Anxiety and depression. A 5-point scale (1) No problems, (2) Slight problems, (3) Moderate problems, (4) Severe problems, and (5) Extreme problems.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 138
score on a scale | 2.1 (0.9) | 2.1 (0.8)

22. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Mobility)
Description: Self-administered questionnaire: Utility-based Health-related Quality of Life - Mobility. A 5-point scale (1) No problems, (2) Slight problems, (3) Moderate problems, (4) Severe problems, and (5) Extreme problems.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 138
score on a scale | 1.5 (0.7) | 1.5 (0.7)

23. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Self-care)
Description: Self-administered questionnaire: Utility-based Health-related Quality of Life - Self-care. A 5-point scale (1) No problems, (2) Slight problems, (3) Moderate problems, (4) Severe problems, and (5) Extreme problems.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 138
score on a scale | 1.1 (0.3) | 1.1 (0.4)

24. Secondary Outcome: Sleep Disturbance T-score
Description: Sleep disturbance T-score, a population scale with a range from 25 (extreme disturbance or impairment) to 80 (not at all) converted from the raw total score of 8-item questionnaire. A score of 50 represents the average of the calibration sample, which was generally more enriched for chronic illness.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 137
score on a scale | 53.4 (9.3) | 55.1 (8.5)

25. Secondary Outcome: Sleep Impairment T-score
Description: Sleep Impairment T-score, a population scale with a range from 25 (extreme disturbance or impairment) to 80 (not at all) converted from the raw total score of 8-item questionnaire. A score of 50 represents the average of the calibration sample, which was generally more enriched for chronic illness.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 132 | 137
score on a scale | 53.4 (9.6) | 55.5 (9.2)

26. Secondary Outcome: Change in Activation of Left Amygdala From Baseline Functional Magnetic Resonance Scan at 2 Months (Regulation of Emotion)
Description: Regulation of emotion, specially activation of the amygdala for nonconscious threat-related emotional reactivity, is assessed using fMRI. In the facial emotion viewing paradigm, facial expression stimuli are standardized black and white photographs of 8 identities (4 female, 4 male) with evoked expressions of threat-related emotions (fear, anger), sad-related emotions (sadness) and reward-related emotions (happiness), along with neutral. To assess amygdala activation for the negative affect circuit, our analysis focused on threatening faces only. Threat stimuli included a combination of fear and anger stimuli relative to neutral blocks. A hemodynamic response convolved boxcar function was used to model the BOLD response for each block of emotional expressions to threat and to sadness relative to neutral face blocks. General linear models were then specified for each task to investigate the contrasts of interest. Higher beta-weight indicates higher activation of the amygdala.
Time Frame: Baseline, 2 months
Population: Not all participants completed fMRI at baseline and 2 months. In addition, quality control diagnostics included removing scans with incidental findings, scanner artefacts, and signal dropout. So the number of participants analyzed is not consistent with the number in the Participant Flow module.
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 35 | 28
beta weights | -0.32 (1.25) | 0.43 (1.69)

27. Secondary Outcome: Change in Activation of Right Amygdala From Baseline Functional Magnetic Resonance Scan at 2 Months (Regulation of Emotion)
Description: as for outcome 26
Time Frame: Baseline, 2 months
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 35 | 28
beta weights | -0.07 (1.38) | 0.01 (0.84)

28. Secondary Outcome: Obesity-related Psychosocial Functioning (Obesity-related Problem Scale)
Description: as for outcome 14
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 127
score on a scale | 51.1 (30.6) | 50.6 (28.6)

29. Secondary Outcome: Anxiety (GAD-7)
Description: as for outcome 15
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 128
score on a scale | 4.8 (4.8) | 5.9 (4.8)

30. Secondary Outcome: Generic Health-related Quality of Life (SF-8 - Physical Component (PCS) )
Description: Self-administered questionnaire - Generic Health-related Quality of Life (SF-8 - physical component (PCS) ). Physical and mental composite scores, a population scale ranged from 0 (lowest quality of life) to 100 (highest quality of life) summed by the total converted scores of each value of the 8 questions. These summary scales have been normalized in the U.S. population (value=50). The higher score indicates better self-reported health-related quality of life.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 127
score on a scale | 47.3 (9.1) | 45.4 (9.3)

31. Secondary Outcome: Generic Health-related Quality of Life (SF-8 - Mental Component (MCS) )
Description: as for outcome 17
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 127
score on a scale | 45.9 (9.9) | 43.9 (9.8)

32. Secondary Outcome: Disability (Sheehan Disability Scale)
Description: as for outcome 18
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 100 | 124
score on a scale | 6 (6) | 6.9 (6.1)

33. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Activity)
Description: as for outcome 19
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 128
score on a scale | 1.5 (0.8) | 1.7 (0.9)

34. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Pain)
Description: as for outcome 20
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 128
score on a scale | 2 (0.8) | 2.3 (0.9)

35. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Anxiety/Depression)
Description: as for outcome 21
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 128
score on a scale | 2 (0.9) | 2.2 (0.9)

36. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Mobility)
Description: as for outcome 22
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 127
score on a scale | 1.6 (0.9) | 1.6 (0.9)

37. Secondary Outcome: Utility-based Health-related Quality of Life (EQ-5D-Self-care)
Description: as for outcome 23
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 128
score on a scale | 1.2 (0.4) | 1.2 (0.5)

38. Secondary Outcome: Sleep Disturbance T-score
Description: as for outcome 24
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 127
score on a scale | 52.9 (9.7) | 55 (8.7)

39. Secondary Outcome: Sleep Impairment T-score
Description: as for outcome 25
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 106 | 127
score on a scale | 52.2 (9.7) | 54.2 (9)

40. Secondary Outcome: Leisure Time Physical Activity
Description: Physical activity was assessed as metabolic equivalent task (MET) minutes per week of leisure-time physical activity of at least moderate intensity based on the sum of the weighted physical activity minutes for moderate (weight: 4 METs), hard (weight: 6 METs), and very hard (weight: 10 METs) activities from the 7-day Physical Activity Recall.
Time Frame: 7-day Physical Activity Recall was administered at 12 months
Population: At 12 months, 169 in RAINBOW intervention and 175 in Usual Care completed the SCL-20, therefore were counted in retention in the Participant Flow module. Among them, 134 in RAINBOW intervention and 139 in Usual care also completed the 7-day Physical Activity Recall at 12 months.
Measure: Mean (Standard Deviation); unit: MET minutes/week
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 134 | 139
MET minutes/week | 704.5 (984.4) | 752.4 (1111.1)

41. Secondary Outcome: Total Energy Expenditure
Description: Totally energy expenditure was measured using the 7-day Physical Activity Recall and provides estimates of total daily energy expenditures (total energy expenditure = sleep hours × 1 MET + light activity hours × 1.5 METs + moderate activity hours × 4 METs + hard activity hours × 6 METs + very hard activity hours × 10 METs).
Time Frame: 7-day Physical Activity Recall was administered at 12 months
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: kilocalories/kilogram/day
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 134 | 139
kilocalories/kilogram/day | 33.1 (2.2) | 33.5 (2.5)

42. Secondary Outcome: Total Calorie Intake
Description: Total calorie intake was measured using 24-hour dietary recalls and provides total energy intake.
Time Frame: One day's 24-hour dietary recall was administered at 12 months
Population: At 12 months, 169 in RAINBOW intervention and 175 in Usual Care completed the SCL-20, therefore were counted in retention in the Participant Flow module. Among them, 131 in RAINBOW intervention and 135 in Usual care also completed the 24-hour diet recalls at 12 months.
Measure: Mean (Standard Deviation); unit: kilocalories/day
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 131 | 135
kilocalories/day | 1592.4 (587.0) | 1591.3 (621.9)

43. Secondary Outcome: DASH (Dietary Approach to Stop Hypertension) Score
Description: Using 24-hour diet recalls, DASH scores were calculated based on combining nine nutrient targets (i.e. total fat, saturated fat, protein, cholesterol, fiber, magnesium, calcium, sodium and potassium). The intermediate target of each nutrient was half-way between the DASH target and population mean (based on the National Health and Nutrition Examination Surveys 2007-2008, latest data available at the inception of the study). For a nutrient, participants reaching the DASH target were assigned one point, those reaching the intermediate target were assigned a half-point, and those not meeting the intermediate target were given 0 points. The DASH score was the sum of points for all nine nutrients and ranged from 0 to 9. DASH score is a measure of diet quality, with higher score indicating higher diet quality
Time Frame: One day's 24-hour dietary recall was administered at 12 months
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAINBOW Intervention Program | Usual Care
Number analyzed (Participants) | 131 | 135
score on a scale | 2.4 (1.3) | 2.5 (1.4)

ADVERSE EVENTS:
Time Frame: Primary and secondary outcome period (up to 24-months)
Arm/Group | RAINBOW Intervention Program | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/205
Serious Adverse Events (participants affected / at risk) | 17/204 | 19/205
Other Adverse Events (participants affected / at risk) | 42/204 | 47/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAINBOW Intervention Program (N=204) | Usual Care (N=205)
Digestive system problem (Gastrointestinal disorders) | 2 (2) | 4 (5)
Diabetes diagnosis (Endocrine disorders) | 0 (0) | 1 (1)
Lymphoma diagnosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Cataract surgery (General disorders) | 0 (0) | 0 (0)
Musculoskeletal problems (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (11) — Adverse Events were monitored in these classifications and cannot be separated.
Nervous system problem (Nervous system disorders) | 0 (0) | 1 (1)
Psychiatric problems (Psychiatric disorders) | 2 (2) | 0 (0)
Reproductive system problems (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Skin problem (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cardiac problems (Cardiac disorders) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAINBOW Intervention Program (N=204) | Usual Care (N=205)
Lymphatic problems (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Cardiac problems (Cardiac disorders) | 3 (3) | 5 (5)
Ear problem (Ear and labyrinth disorders) | 0 (0) | 0 (0)
Endocrine problems (Endocrine disorders) | 1 (1) | 1 (1)
Digestive system problem (Gastrointestinal disorders) | 5 (6) | 8 (9)
Other problems (General disorders) | 0 (0) | 0 (0)
Musculoskeletal problems (Musculoskeletal and connective tissue disorders) | 22 (30) | 24 (30) — Adverse Events were monitored in these classifications and cannot be separated.
Benign tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Nervous system problem (Nervous system disorders) | 5 (5) | 6 (11)
Psychiatric problem (Psychiatric disorders) | 1 (1) | 1 (1)
Reproductive system problems (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Respiratory problem (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 5 (7)
Skin problems (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8)
Vascular problems (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02246413/Prot_SAP_000.pdf